CLINICAL TRIAL: NCT04891965
Title: A Randomized, Placebo-Controlled, Double-Blind, Phase 1 Study of ART24 in Subjects Recently Cured of a Clostridioides Difficile Infection (CDI)
Brief Title: A Study of ART24 in Subjects Recently Cured of a Clostridioides Difficile Infection (CDI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adiso Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ART24-1-001
Record Dates: First submitted 2021-04-29; First posted 2021-05-19 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Clostridium Difficile Infection Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ART24 (Cohort A) (Experimental): In Cohort A, subjects will receive ART24 or placebo daily for 7 days
  Interventions: Biological: ART24
- Placebo (Cohort A) (Placebo Comparator): In Cohort A, subjects will receive ART24 or placebo daily for 7 days
  Interventions: Drug: Placebo
- ART24 (Cohort B) (Experimental): In Cohort B, subjects will receive ART24 or placebo daily for 28 days
  Interventions: Biological: ART24
- Placebo (Cohort B) (Placebo Comparator): In Cohort B, subjects will receive ART24 or placebo daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ART24 — Each ART24 capsule will contain lyophilized ART24 and inactive excipients. ART24 will be supplied in a dose strength of 5×10^9 CFU/capsule. Subjects will receive 1 capsule daily.
  Other Names: ADS024
  Arms: ART24 (Cohort A); ART24 (Cohort B)
Drug: Placebo — Each placebo capsule is identical in appearance, weight, and packaging to ART24 capsules, but will contain only the inactive excipients. Subjects will receive 1 capsule daily.
  Arms: Placebo (Cohort A); Placebo (Cohort B)

SUMMARY:
This is a randomized, placebo-controlled, double-blind, multi-site study in which up to approximately 36 subjects with a recent C. difficile infection (CDI) who have completed a standard of care course of CDI antibiotics and have achieved clinical cure based on signs and symptoms, will be randomized to 7 or 28 daily doses of ART24 or placebo. Subjects will be followed for 6 months after the last dose of study drug.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, multi-site study in which up to approximately 36 subjects with a recent CDI (primary [meaning the first occurrence they have had] or recurrent infection) who have completed a standard of care course of CDI antibiotics (vancomycin, fidaxomicin, or metronidazole administered for 10 to 21 days) and have achieved clinical cure based on signs and symptoms, will be randomized to 7 or 28 daily doses of ART24 or placebo. Subjects will be followed for 6 months after the last dose of study drug.

Subjects will receive study drug in the following 2 sequential cohorts:

* Cohort A: ART24 or placebo once daily for 7 days (8 subjects)
* Cohort B: ART24 or placebo once daily for 28 days (28 subjects)

In each cohort, subjects will be randomized in a ratio of 3 [active]:1 [placebo]. Subjects who are randomized to active treatment in both cohorts will receive ART24 (5×10^9 colony-forming units [CFU]) daily.

Initiation of Cohort B will only occur once the Data Review Committee (DRC) has evaluated blinded safety data (through Week 2) from Cohort A and recommends that the study proceed to the next cohort.

ELIGIBILITY:
Inclusion Criteria:

* Have successfully completed a full course of a standard of care CDI antibiotic for a qualifying CDI episode (primary or recurrent) within 3 to 7 days of randomization

  * Qualifying CDI episode must meet all of the following (3) criteria

    1. Positive stool C. difficile toxin (NAAT, EIA, CCTA, or equivalent test) as documented by study site AND
    2. History of ≥3 unformed stools (Bristol scores of 5, 6, or 7) within 24 hours
    3. Received standard of care antibiotic treatment for CDI diagnosis
* Prior to the first dose of study drug, completion of standard of care antibiotic therapy with oral vancomycin, metronidazole, or fidaxomicin for CDI with a treatment duration of 10 to 21 days
* Clinical cure assessed at Day 1 visit (randomization) defined as ≤2 unformed stools per day for at least 2 consecutive days and maintained through Day 1 without the need for further antibiotic therapy
* Able to begin treatment with study drug within 3 to 7 days following completion (i.e., last dose) of the CDI antibiotic course for the qualifying CDI episode

Exclusion Criteria:

* Body mass index ≥40.0 kg/m2
* Life expectancy of ≤12 months
* Inpatient (in hospital or skilled nursing facility) at the time of randomization
* Current (i.e., qualifying) CDI episode required admission to an Intensive Care Unit
* Pregnant, breastfeeding, or seeking pregnancy while on study
* Have, as determined by the Investigator, a history or clinical/laboratory manifestations of significant neurological, renal, hepatic, hematologic, cardiac, pulmonary, metabolic, endocrine, psychiatric, GI disorders other than CDI (including infectious, ischemic, or immunological diseases), human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV) infection, or other condition that could interfere with the evaluation of safety or efficacy, or put the subject at risk of harm from study participation
* Have an active malignancy of any type or history of a malignancy within past 5 years, except for treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Have an acute febrile illness (fever >38°C [100.4°F]) at Day 1
* Drug, alcohol, or substance dependence within the last 2 years
* Any of the following laboratory results at Screening:

  * White blood cell count ≥15,000 cells/mm3
  * Absolute neutrophil count <1000/mm3
  * Liver function test result (e.g., aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), or total bilirubin) of ≥3 times the upper limit of normal
  * Serum albumin <3 g/dL
  * Serum creatinine >1.8 mg/dL and oliguric
* Use of systemic antibiotic therapy for conditions other than CDI within 7 days of randomization or expectation to require antibiotic therapy for conditions other than CDI for 12 weeks following the first dose of study drug for Cohort A or 16 weeks following the first dose of study drug for Cohort B, including subtherapeutic doses of oral antibiotics (e.g., for rosacea)
* Have a known immunodeficiency disorder, including but not limited to:

  * An immunodeficiency disease
  * Receiving, or plans to receive, treatment with systemic corticosteroids equivalent to >10 mg prednisone per day
  * Receiving, or plans to receive, myelosuppressive chemotherapy
* Previous fecal transplant or live biotherapeutic product within 1 year of randomization
* Treatment with bezlotoxumab (Zinplava™) for the qualifying CDI episode
* Diagnosis of inflammatory bowel disease (including but not limited to: Crohn's disease, ulcerative colitis, microscopic colitis)
* Active irritable bowel syndrome [those with diarrhea predominant or alternating constipation and diarrhea] (in past 6 months based on Rome IV criteria and subject deemed not suitable for study by Investigator's judgment)
* Celiac disease not well controlled on gluten-free diet
* Active gastroparesis, toxic megacolon, pseudomembranous colitis, colostomy, intestinal resection (except appendectomy), ileus or short gut syndrome
* History of chronic diarrhea apart from prior CDI
* Intra-abdominal surgery, including laparoscopic procedures, within 8 weeks of Screening (appendectomy and cholecystectomy excluded)
* History of difficulty swallowing food or liquids
* Taking antidiarrheal agents (e.g., loperamide) or laxatives (e.g., senna) on a regular basis
* Use of non-dietary probiotic supplements within 7 days of Day 1 or plan to use non-dietary probiotic supplements while on study through Week 12 in Cohort A and Week 16 in Cohort B
* Known to have consumed fermented or other foods that may contain B. amyloliquefaciens (such as miso, soybean paste, or fermented rice- or locust bean-derived products) within 7 days prior to Day 1, or plan to consume them prior to Week 12 for Cohort A and prior to Week 16 for Cohort B
* Participation in a clinical trial of an investigational drug or medical device within 30 days or 5 half-lives, whichever is longer, prior to the Screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of ART24 based on the percentage of subjects experiencing treatment-emergent adverse events (TEAEs). | Randomization through the week 12 study visit (Cohort A) or week 16 study visit (Cohort B)
  The percentage of subjects experiencing a TEAE will be summarized using the MedDRA system organ class and preferred term.
Assess the safety and tolerability of ART24 based on the number of subjects observed with a change from baseline in clinical laboratory tests, vital signs, physical examination. | Randomization through the week 12 study visit (Cohort A) or week 16 study visit (Cohort B)
  The number of subjects with a change from baseline from normal to abnormal in clinical laboratory test results, vital signs, physical examination will be summarized.

SECONDARY OUTCOMES:
Recurrence of CDI | Randomization through the week 12 study visit (Cohort A) or week 16 study visit (Cohort B)
  Defined as ≥3 unformed stools (Bristol Scores of 5, 6, or 7) within 24 hours, AND positive stool testing for C. difficile toxin as documented by the central laboratory, AND the need for antibiotic retreatment for CDI diagnosis.
Time to CDI Recurrence | Through the week 12 study visit (Cohort A) or week 16 study visit (Cohort B)
  Evaluating the time to CDI recurrence (if applicable) relative to the administration of study medication
Hospitalization for CDI | Randomization through the week 12 study visit (Cohort A) or week 16 study visit (Cohort B)
  Evaluating the proportion of subjects who are hospitalized due to a CDI recurrence
ART24-positive Fecal Samples | Randomization through the week 12 study visit (Cohort A) or week 16 study visit (Cohort B)
  Proportion of subjects with ART24-positive fecal sample assessed at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Renu Gupta, MD, Study Director — Adiso Therapeutics, Inc.
Locations (15):
- United States (13):
  - Palmtree Clinical Research, Palm Springs, California
  - Gastro Florida, Clearwater, Florida
  - Doral Medical Research, Doral, Florida
  - Louisiana Research Center, Shreveport, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Mercury Street Medical Group, Butte, Montana
  - DiGiovanna Institute, Massapequa, New York
  - NYU Grossman School of Medicine, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Advanced Clinical Research, Riverton, Utah
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - Intermed Groupe Sante, Chicoutimi, Quebec

IPD SHARING:
Plan to Share IPD: No